CLINICAL TRIAL: NCT02486562
Title: IConquerMS™ - a Patient-Powered Research Network for Multiple Sclerosis
Acronym: iCMS
Status: Recruiting | Type: Observational
Sponsor: Accelerated Cure Project for Multiple Sclerosis (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Ogilvy (Unknown); Arizona State University (Other)
Responsible Party: Sponsor
Other Study IDs: ACP-MS-PPRN-001
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People diagnosed with Multiple Sclerosis

SUMMARY:
iConquerMS™ is a research initiative developed by and for people with multiple sclerosis (MS) to contribute their health data and ideas to advance and accelerate research into MS. iConquerMS welcomes adults with MS and others interested in advancing MS research, children and teens with MS and their family members (via iConquerMS Kids & Teens) and MS caregivers (via iConquerMS Caregivers) to participate.

DETAILED DESCRIPTION:
The purpose of this study is to create a Multiple Sclerosis Patient-Powered Research Network (MS-PPRN) that includes at least 20,000 people with multiple sclerosis (MS) who contribute data on their health and other topics. Survey data will be made available to research scientists who are studying MS and similar diseases. Our goal is to use this data to answer questions that researchers and people with MS have regarding the disease, including its causes, treatments, and other topics.

While the MS-PPRN is focused on enrolling people with MS, people without MS are also welcome to participate in this research study. Adults are invited to participate via iConquerMS, while children and teens are invited to participate via iConquerMS Kids & Teens. Adults who are MS caregivers may participate via the dedicated iConquerMS Caregivers site.

This study will be conducted online via the iConquerMS.org website. This is an ongoing study and will last for an indefinite period of time.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older at the time of informed consent or under 21 with parental consent and participant assent.

Exclusion Criteria:

* Unwilling or unable to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary cohort is people with multiple sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2014-11; Primary Completion 2030-10 (Estimated); Study Completion 2036-10 (Estimated)

PRIMARY OUTCOMES:
Number of people with multiple sclerosis who experience health-related quality-of-life changes | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Accelerated Cure Project, Waltham, Massachusetts, United States